CLINICAL TRIAL: NCT03887689
Title: Early Psychological Intervention After Rape: a Feasibility Study
Brief Title: Early Psychological Intervention After Rape
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, Principal investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016/2194-31
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified prolonged exposure (Experimental): Participants will receive three sessions of modified prolonged exposure therapy.
  Interventions: Behavioral: Modified prolonged exposure

INTERVENTIONS:
Behavioral: Modified prolonged exposure — Participants will receive three sessions of modified prolonged exposure therapy.

SUMMARY:
The aim of the study is to translate and adapt a brief treatment protocol based on prolonged exposure provided within 72 hours after a rape to a Swedish context and pilot test feasibility and delivery in ten executive patients recruited at the Emergency Clinic for Rape victims in Stockholm.

DETAILED DESCRIPTION:
The aim of the study is to translate and adapt a brief treatment protocol based on prolonged exposure provided within 72 hours after a rape to a Swedish context and pilot test feasibility and delivery in ten executive patients recruited at the Emergency Clinic for Rape victims in Stockholm.

ENDPOINTS The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), Beck Depression Inventory (BDI) at baseline and post-treatment.

Insomnia Severity Index (ISI) , Multidimensional Scale of Perceived Social Support (MSPSS), World Health Organization Disability Assessment Schedule(WHODAS-12) at post-treatment.The clinician-administered PTSD scale for DSM-5 (CAPS-5) at follow up.

Data on feasibility aspects of the intervention will also be collected: compliance to the intervention/homework/assessments, possibilities to recruit, adverse events.

Recruitment The investigatorors will recruit ten consecutive patients attending at the Emergency Clinic for Rape victims at Stockholm South Hospital, Sweden.

Safety parameters Participants had the opportunity to report any adverse events during treatment, at posttreatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Attending at the Emergency Clinic for Rape victims at Stockholm South Hospital, Sweden within 72 hours after experiencing a rape)
* Remembered the event.

Exclusion Criteria:

* ongoing suicidal ideation or attempted suicide within the last two months
* ongoing self-harm behavior
* ongoing intoxication
* other serious psychiatric comorbidity (ongoing psychotic symptoms or manic episode)
* low cognitive capacity
* not fluent in Swedish
* subjected to ongoing violence or threat

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
CLINICIAN-ADMINISTERED PTSD SCALE for Diagnostic and Statistical Manual of Mental Disorders-5 (CAPS) | Change 2 months (primary endpoint) after intervention
  Clinical interview that gives a continuous measure of PTSD severity and dichotomous diagnosis of PTSD

SECONDARY OUTCOMES:
PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-5 (PCL-5) | Change 2 months after intervention
  Change in symptoms of post traumatic stress from post treatment and follow up (2 months). The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. All items are scored on a 0-4 scale. Higher score indicate worse severity.
Beck Depression Inventory (BDI) | Change 2 months after intervention
  Change in depressive symptoms from baseline to post treatment and follow up (2 months). The BDI is a 21 item self-report measure that assesses the presence and severity of depressive symptoms. All items are scored on a 0-3 scale. Higher score indicate worse severity.
Adverse Events | Change 2 months after intervention
  Number of adverse events from baseline to follow up 2 months
WHO Disability Assessment Schedule (WHODAS) | Change 2 months after intervention
  Measure of general health and function. The WHODAS-12 is a 12 item self-report measure that assesses overall health and functioning. All items are scored on a 0-4 scale. Higher score indicate worse severity.
Insomnia Severity Index (ISI) | Change 2 months after intervention
  Self-report questionnaire regarding insomnia. The ISI is a 12 item self-report measure that assesses sleep quality. All items are scored on a 0-4 scale. Higher score indicate worse severity.
Multidimensional Scale of Perceived Social Support (MSPSS) | Change 2 months after intervention
  A measure to assess for social support. MSPSS is a 7 item self-report measure that assesses aspects of social support. All items are scored on a 0-7 scale. Lower score indicate worse severity.
Intrusion diary | Change at week 1, week 2 and week 3 of the intervention.
  Change in self-report assessment of daily intrusions using a pen and stencil diary.

IPD SHARING:
Plan to Share IPD: No